CLINICAL TRIAL: NCT02634879
Title: Behavioral Economics in Provider Incentive Design
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Amol Navathe, Principal Investigator, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 823358
Record Dates: First submitted 2015-12-07; First posted 2015-12-18 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Control Group
- Loss Aversion (Active Comparator): Each physician in this arm will have access to funds prior to earning them.
  Interventions: Behavioral: Incentive Change
- Group Incentive (Active Comparator): Each physician will receive 50% of their potential incentive based on group performance. Physicians will also receive information on the performance of physicians on key CI measures in their group.
  Interventions: Behavioral: Incentive Change

INTERVENTIONS:
Behavioral: Incentive Change
  Arms: Group Incentive; Loss Aversion

SUMMARY:
The shift towards value-based reimbursement in U.S. healthcare is accelerating. Payment reform initiatives have taken many shapes-accountable care organizations, bundled payments, value-based purchasing, medical homes, global payment-but all share the common strategy of tying provider (physician, hospital, health system) reimbursement to performance on costs, outcomes, or both. Yet, pay-for-performance has demonstrated little effect on physician behavior and patient outcomes. Payers and provider groups are in need of novel approaches to structure provider incentives-both financial and non-financial-to better promote the delivery of quality, cost-effective care. In this project, the study team plans to study how behavioral economic principles can improve the effectiveness of physician incentives to deliver higher quality and lower cost care. They will test the application of specific behavioral economic principles including immediacy, social pressure, and loss aversion in incentive design and implementation. The study will contribute to an empirical foundation for re-design of existing physician incentive programs and implementation of new policies through secondary data analyses and a multi-arm experiment that evaluate the impact of promising behavioral economics principles on the effectiveness of provider financial and nonfinancial incentives.

DETAILED DESCRIPTION:
The key goal of this project is to demonstrate how using behavioral economic principles to inform the structure of provider incentives and the practice environment can improve provider performance, especially in settings that are moving away from fee-for-service reimbursement and fragmented care towards new payment and delivery models that emphasize coordination of care and provider accountability. The project will build upon the recently completed 'Phase 1' project in which a set of behavioral economic approaches to provider performance were identified that could meaningfully improve provider performance, a focused research agenda of high-priority tests of these concepts (i.e., content of this proposal) was developed; and information on how behavioral economics can be used to improve incentives for physicians was disseminated. For this phase, an experimental evaluation will be conducted of the impact of social pressure by varying individual and group incentives and the comparative effectiveness of two loss aversion framing methods (endowment versus performance gap) on provider performance via a multi-arm experiment. We will complement the quantitative evaluations with pre- and post-intervention qualitative surveys of physicians and patients to better understand the influence on behavior change, culture, acceptability of the incentive program, and patient reported outcomes on health and experience.

ELIGIBILITY:
Inclusion Criteria:

* Physician at participating provider organization (PCP and specific specialties)

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2016-01; Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Physician performance | Baseline to 12 months
  Measured by physician-level CI composite quality measure score

SECONDARY OUTCOMES:
Physician Practice Behavior | Baseline to 12 months
  Evaluate how practice behavior changes by looking at pre and post survey data.
Physician Incentive Payouts | Throughout the 12 months
  How much incentives the physicians receive throughout the project.
Patient satisfaction | 6 months to 12 months
  Patients will be surveyed to assess their satisfaction with their physician throughout the project period.

CONTACTS AND LOCATIONS:
Overall Officials: Amol Navathe, MD, PhD, Principal Investigator — University of Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Navathe AS, Volpp KG, Caldarella KL, Bond A, Troxel AB, Zhu J, Matloubieh S, Lyon Z, Mishra Meza A, Sacks L, Nelson C, Patel P, Shea J, Calcagno D, Vittore S, Sokol K, Weng K, McDowald N, Crawford P, Small D, Emanuel EJ. Effect of Financial Bonus Size, Loss Aversion, and Increased Social Pressure on Physician Pay-for-Performance: A Randomized Clinical Trial and Cohort Study. JAMA Netw Open. 2019 Feb 1;2(2):e187950. doi: 10.1001/jamanetworkopen.2018.7950. PMID 30735234